CLINICAL TRIAL: NCT01487148
Title: POCARED Diagnostics, LTD, Field Study Protocol
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Pocared Diagnostics (Industry)
Responsible Party: Sponsor
Other Study IDs: POCARED001
Record Dates: First submitted 2011-12-02; First posted 2011-12-07 (Estimated); Last update posted 2011-12-07 (Estimated); Status verified 2011-12

CONDITIONS: Urinary Tract Infections
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: None Retained — Samples are de-identified leftover samples.
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is designed to compare the performance of the P-1000 System, POCARED's Rapid Diagnostic System which uses optical fluorescence analysis, to standard methods of uropathogen quantification and identification.

DETAILED DESCRIPTION:
This study will be conducted at 5 sites, 4 in the United States and 1 site in Israel. 40,000 clinical specimens will be included and assessed by the laboratories using standard reference methods and the P-1000.

ELIGIBILITY:
Inclusion Criteria:

* Samples arriving in the laboratory for urine culture

Exclusion Criteria:

* Samples <=2mL
* Specimens stored at room temperature for more than 2 hours (unless a preservative is used)
* Specimens refrigerated for more than 24 hours
* Specimens requesting low count urine culture (<100,000 CFU/mL [colony forming units per milliliter])
* Bloody specimens

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: At least 70 consecutive leftover and de-identified urine samples arriving in the laboratory each day for culture will be tested.
Sampling Method: Non-Probability Sample
Enrollment: 40000 (Estimated)
Dates: Start 2011-12; Primary Completion 2012-06 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Agreement | 6 months
  Agreement of the POCARED quantification and identification compared with standard methods.
Sensitivity | 6 months
  Sensitivity of the POCARED quantification and identification compared with standard methods.
Specificity | 6 months
  Specificity of the POCARED quantification and identification compared with standard methods.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Gurfinkel, Study Director — POCARED Diagnostics, Ltd.
Locations (5):
- United States (4):
  - Southern California Permanente Medical Group (SCPMG) Regional Reference Laboratories, North Hollywood, California
  - Mayo Clinic, Rochester, Minnesota
  - Cleveland Clinic, Cleveland, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
- Chaim Sheba Medical Center, Tel Aviv, Israel